CLINICAL TRIAL: NCT02271945
Title: A Phase 1b/2 Open-label Study to Evaluate the Safety/Efficacy of MEDI-551 in Combination With Immunomodulating Therapy in Subjects With Relapsed or Refractory Aggressive B-cell Lymphomas
Brief Title: Safety/Efficacy of MEDI-551 in Combination With Immunomodulating Therapies in Subjects With Aggressive B-cell Lymphomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D2852C00004
Record Dates: First submitted 2014-09-23; First posted 2014-10-22 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Relapsed/Refractory Aggressive B-cell Lymphomas
Keywords: aggressive lymphoma, DLBCL, NHL
MeSH Terms: conditions — Recurrence; Lymphoma, Non-Hodgkin | interventions — inebilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg (Experimental): Participants will receive intravenous (IV) infusion of MEDI-551 12 mg/kg on Days 1 and 8 of Cycle 1 and Day 1 of Cycle 2 through Cycle 13 (each cycle of 28 days) and IV infusion of MEDI0680 2.5 mg/kg on Days 2 and 15 of Cycle 1 and Days 1 and 15 of Cycle 2 through Cycle 13.
  Interventions: Drug: MEDI-551 12 mg/kg; Drug: MEDI0680 2.5 mg/kg
- MEDI-551 12 mg/kg and MEDI0680 10 mg/kg (Experimental): Participants will receive IV infusion of MEDI-551 12 mg/kg on Days 1 and 8 of Cycle 1 and Day 1 of Cycle 2 through Cycle 13 (each cycle of 28 days) and IV infusion of MEDI0680 10 mg/kg on Days 2 and 15 of Cycle 1 and Days 1 and 15 of Cycle 2 through Cycle 13.
  Interventions: Drug: MEDI-551 12 mg/kg; Drug: MEDI0680 10 mg/kg

INTERVENTIONS:
Drug: MEDI-551 12 mg/kg — Participants will receive intravenous (IV) infusion of MEDI-551 12 mg/kg on Days 1 and 8 of Cycle 1 and Day 1 of Cycle 2 through Cycle 13
Drug: MEDI0680 2.5 mg/kg — Participants will receive IV infusion of MEDI0680 2.5 mg/kg on Days 2 and 15 of Cycle 1 and Days 1 and 15 of Cycle 2 through Cycle 13.
  Arms: MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg
Drug: MEDI0680 10 mg/kg — Participants will receive IV infusion of MEDI0680 10 mg/kg on Days 2 and 15 of Cycle 1 and Days 1 and 15 of Cycle 2 through Cycle 13.
  Arms: MEDI-551 12 mg/kg and MEDI0680 10 mg/kg

SUMMARY:
This is a Phase 1b/2 open-label study to evaluate the safety/efficacy of MEDI-551 + MEDI0680 in participants with relapsed or refractory aggressive B-cell lymphomas who have failed 1-2 prior lines of therapy.

DETAILED DESCRIPTION:
This is a Phase 1b/2, multicenter, open-label, study of MEDI-551 in combination with immunomodulating therapy evaluating the safety, tolerability, pharmacokinetics, immunogenicity and anti-tumor activity in subjects with relapsed or refractory aggressive B-cell lymphomas

ELIGIBILITY:
Key inclusion criteria:

* Histologically confirmed aggressive diffuse large B-cell lymphoma (DLBCL), including follicular lymphoma (FL) transforming to DLBCL, transformed indolent lymphoma, mantle cell lymphoma (MCL), or Grade 3B FL for dose-escalation cohorts. Only participants with DLBCL will be enrolled in the dose-expansion cohort.
* Willing to provide a fresh tumor sample
* Evaluable/measurable disease with measurable disease defined as greater than or equal to (>= 1) lesion less than or equal to (<=) 20 mm in one dimension or ≥ 15 mm in 2 dimensions as measured by conventional or high-resolution (spiral) computed tomography (CT). Disease evaluable by the International Working Group criteria (Cheson et al, 2007). (NOTE: Irradiated lesions will not be evaluable.)
* Baseline fludeoxyglucose positron emission tomography (FDG-PET) or FDG-PET/CT scans must show positive lesions compatible with CT-defined anatomical tumor sites.
* Relapsed from or refractory to >= 2 prior chemotherapy regimens with >= 1 regimen containing rituximab or failed 1 prior rituximab-containing regimen and unable to tolerate additional multiagent chemotherapy. NOTE: Subjects enrolled in the dose-escalation portion of the study must have exhausted all available standard therapy.
* At least 100 days past autologous stem cell transplant (ASCT).
* At least 1 year past allogeneic stem-cell transplant (SCT) and off immunosuppression therapy, with no evidence of graft-versus-host disease.
* Eastern Cooperative Oncology Group performance status 0-2.
* Adequate hematological function
* Adequate organ function
* Females of childbearing potential who are sexually active with a nonsterilized male partner must use a highly effective method of contraception for 30 days prior to the first dose of investigational product, and must agree to continue using such precautions for 180 days after the final dose of investigational product.
* Nonsterilized males who are sexually active with a female partner of childbearing potential must use a highly effective method of contraception from Day 1through 90 days after receipt of the final dose of investigational product.

Key exclusion criteria:

* Any concurrent chemotherapy, radiotherapy, immunotherapy, biologic or hormonal therapy for treatment of cancer.
* Receipt of any experimental therapy, mAb, cancer vaccine, chemotherapy or small molecule within 28 days prior to Cycle 1 Day 1 or 5 half-lives of that therapy, whichever is shorter.
* Previous therapy directed against cluster of differentiation 19 (CD19)
* Prior exposure to immunotherapy such as but not limited to other anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4), anti-PD 1, or anti-PD-L1 antibodies excluding cancer vaccines.
* Vaccination with a live virus within 28 days prior to receiving the first dose of study drug
* History of other invasive malignancy within 2 years except for cervical carcinoma in situ, non-melanomatous carcinoma of the skin or ductal carcinoma in situ of the breast that has been surgically cured.
* Evidence of significant active infection requiring antimicrobial, antifungal, antiparasitic, or antiviral therapy or for which other supportive care is given unless the subject is clinically stable.
* Human immunodeficiency virus (HIV) positive serology or acquired immunodeficiency syndrome (AIDS).
* Active hepatitis B
* Ongoing >= Grade 2 toxicities from previous cancer therapies or any unresolved > Grade 1 immune-related adverse event (irAE) event unless specifically allowed in the inclusion/exclusion criteria.
* No immunosuppressive therapy within 14 days of Cycle 1 Day 1 of MEDI0680 (AMP-514) dosing.
* Active or prior documented autoimmune or inflammatory disease except vitiligo.
* History of primary immunodeficiency.
* Major surgical procedures (as defined by the principal investigator) within 28 days of Cycle 1 Day 1 or still recovering from prior surgery.
* History of tuberculosis, including those who may have completed prophylactic isoniazid (INH) therapy.
* Documented current central nervous system (CNS) involvement, leptomeningeal disease, or spinal cord compression.
* Pregnancy or lactation.
* Clinically significant abnormality on electrocardiogram (ECG).
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, current pneumonitis, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs from MEDI-551 or MEDI0680 (AMP-514), or compromise the ability of the subject to give written informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-05-24 (Actual); Study Completion 2016-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (6):
- United States (6):
  - Research Site, Birmingham, Alabama
  - Research Site, Baltimore, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, The Bronx, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 01Dec2014 to 24May2016.
Pre-assignment Details: A total of 16 participants were screened in this study. Of which, 6 participants failed screening and 10 participants were enrolled in the study and received the study drugs.
Groups:
- MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg: Participants received IV infusion of MEDI-551 12 mg/kg on Days 1 and 8 of Cycle 1 and Day 1 of Cycle 2 through Cycle 13 (each cycle of 28 days) and IV infusion of MEDI0680 2.5 mg/kg on Days 2 and 15 of Cycle 1 and Days 1 and 15 of Cycle 2 through Cycle 13.
- MEDI-551 12 mg/kg and MEDI0680 10 mg/kg: Participants received IV infusion of MEDI-551 12 mg/kg on Days 1 and 8 of Cycle 1 and Day 1 of Cycle 2 through Cycle 13 (each cycle of 28 days) and IV infusion of MEDI0680 10 mg/kg on Days 2 and 15 of Cycle 1 and Days 1 and 15 of Cycle 2 through Cycle 13.
Period: Overall Study
Arm/Group | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg
Started | 5 | 5
Completed | 0 | 0
Not Completed | 5 | 5
Not completed — Death | 3 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- TOTAL: Total of all reporting groups
Arm/Group | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg | TOTAL
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 63.2 (7.1) | 63.8 (14.8) | 63.5 (11.0)
Age, Customized [Count of Participants; unit: Participants]
  < 65 YEARS | 3 | 3 | 6
  >= 65 YEARS | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Data for the participants in the category for "Other" is included under "unknown or not reported" category.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 4 | 4 | 8
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of MEDI-551
Description: The Maximum Tolerated Dose, defined as the highest dose where less than or equal to (<= 1) out of 6 subjects experiences a dose limiting toxicity (DLT) during the DLT evaluation period (Day 1 to Day 28 of Cycle 1) or the highest protocol specified dose not exceeding MTD.
Time Frame: Day 1 to Day 28 of Cycle 1 (28-day cycle)
Population: Evaluable Population for DLT included all participants in the dose escalation portion who received all protocol assigned doses and completed safety follow-up during the first 28-day period of therapy, or experienced a DLT during the DLT evaluation period.
Measure: Number; unit: mg/kg
Arm/Group | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg
Number analyzed (Participants) | 3 | 4
mg/kg | NA — The study was terminated before the MTD was reached. | NA — The study was terminated before the MTD was reached.

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) or Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An Adverse Event (AE) is any unfavourable and unintended signs, symptoms, or diseases temporally associated with use of study drug, whether or not considered related to study drug. SAE is any AE that resulted in death, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, life-threatening, a congenital anomaly/birth defect, or an important medical event. TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug, up to 90 days after the end of treatment (EOT).
Time Frame: From treatment administration to 90-days after last dose of study drug (up to approximately 2 years)
Population: As-treated Population included all participants who were treated with study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg
Number analyzed (Participants) | 5 | 5
Participants
  TEAEs | 5 | 5
  TESAEs | 2 | 1

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Related to Clinical Laboratory Abnormalities
Description: An abnormal laboratory findings that was judged by the investigator to be medically significant was reported as an AE. TEAEs were defined as events present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug, for the period extending to 90 days after the end of study drug.
Time Frame: From treatment administration to 90-days after last dose of study drug (up to approximately 2 years)
Population: As-treated Population included all participants who were treated with study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg
Number analyzed (Participants) | 5 | 5
Participants
  Febrile neutropenia | 1 | 0
  Hypoglobulinaemia | 0 | 1
  Blood alkaline phosphatase increased | 0 | 1
  Blood creatinine increased | 1 | 0
  Blood pressure increased | 1 | 0
  Lymphocyte count decreased | 0 | 2
  Neutrophil count decreased | 0 | 1
  Platelet count decreased | 0 | 1
  White blood cell count decreased | 0 | 1
  Hyperglycaemia | 0 | 2
  Hyperuricaemia | 1 | 0
  Hypocalcaemia | 0 | 1
  Hyponatraemia | 0 | 1
  Haematuria | 1 | 0
  Proteinuria | 0 | 1

4. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Related to Vital Signs, Physical Findings Abnormalities
Description: Vital signs included parameters such as blood pressure, temperature, respiratory rate, and pulse oximetry. An abnormal vital signs and physical findings that was judged by the investigator to be medically significant was reported an AE. TEAEs were defined as events present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug, for the period extending to 90 days after the end of study treatment.
Time Frame: From treatment administration to 90-days after last dose of study drug (up to approximately 2 years)
Population: As-treated Population included all participants who were treated with study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg
Number analyzed (Participants) | 5 | 5
Participants
  Infusion related reaction | 1 | 2
  Pyrexia | 0 | 1

5. Primary Outcome: Number of Participants With Best Overall Response
Description: The best overall response was calculated, based upon the disease assessments recorded during the study visits, and summarized with the number of participants for the following categories: complete response (disappearance of all evidence of disease), partial response (regression of measurable disease and no new sites), stable disease (SD), progessive disease (PD), and non- evaluable (NE).
Time Frame: Day 1 to Day 28 of Cycle 13 (28-day cycle)
Population: As-treated Population included all participants who were treated with study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg
Number analyzed (Participants) | 5 | 5
Participants
  Complete Response | 0 | 1
  Partial Response | 0 | 0
  Stable Disease | 0 | 1
  Progressive Disease | 5 | 3
  Non-evaluable | 0 | 0

6. Secondary Outcome: Mean Peak and Trough Concentrations of MEDI551
Description: The mean peak and Trough concentration of MEDI551 were observed. Peak is the end of infusion measurement and the Trough is the pre-dose measurement.
Time Frame: End of Infusion (EOI) of Cycle 1 Day 1; Pre-dose and EOI of C1D8, C2D1, C3D1 and C4D1
Population: As-treated Population included all participants who were treated with study drug.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg
Number analyzed (Participants) | 5 | 5
mcg/mL
  Cycle1 Day1 End of Infusion | 244 (49.3) | 220 (66.2)
  C1D8 Predose | 103 (13.3) | 96.8 (38.3)
  C1D8 End of Infusion | 329 (63.4) | 313 (74.2)
  C2D1 Predose: number analyzed (Participants) | 2 | 4
  C2D1 Predose | 92.4 (36.3) | 103 (45.4)
  C2D1 End of Infusion: number analyzed (Participants) | 2 | 3
  C2D1 End of Infusion | 276 (59.1) | 336 (76.1)
  C3D1 Predose: number analyzed (Participants) | 2 | 3
  C3D1 Predose | 109 (26.8) | 108 (49.9)
  C3D1 End of Infusion: number analyzed (Participants) | 2 | 2
  C3D1 End of Infusion | 325 (71.8) | 300 (55.2)
  C4D1 Predose: number analyzed (Participants) | 1 | 2
  C4D1 Predose | 85.7 (NA) — Standard Deviation was not evaluable as insufficient number of participants. | 111 (57.2)
  C4D1 End of Infusion: number analyzed (Participants) | 1 | 2
  C4D1 End of Infusion | 338 (NA) — Standard Deviation was not evaluable as insufficient number of participants. | 292 (77.8)

7. Secondary Outcome: Mean Peak and Trough Concentrations of MEDI0680
Description: The mean peak and Trough concentration of MEDI0680 were observed. Peak is the end of infusion measurement and the Trough is the pre-dose measurement.
Time Frame: EOI of Cycle 1 Day 2; Pre-dose and EOI of C1D15, C2D1, C3D1 and C4D1
Population: As-treated Population included all participants who were treated with study drug.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg
Number analyzed (Participants) | 5 | 5
mcg/mL
  C1D2 End of Infusion: number analyzed (Participants) | 5 | 4
  C1D2 End of Infusion | 49.8 (18.2) | 256 (101)
  C1D15 Predose | 18.7 (2.10) | 109 (30.1)
  C1D15 End of Infusion: number analyzed (Participants) | 4 | 5
  C1D15 End of Infusion | 72.5 (12.4) | 298 (41.7)
  C2D1 Predose: number analyzed (Participants) | 3 | 3
  C2D1 Predose | 32.8 (6.31) | 178 (52.3)
  C2D1 End of Infusion: number analyzed (Participants) | 2 | 2
  C2D1 End of Infusion | 92.9 (17.1) | 339 (55.9)
  C3D1 Predose: number analyzed (Participants) | 2 | 3
  C3D1 Predose | 44.1 (3.25) | 277 (64.3)
  C3D1 End of Infusion: number analyzed (Participants) | 2 | 1
  C3D1 End of Infusion | 110 (29.6) | 590 (NA) — Standard Deviation was not evaluable as insufficient number of participants.
  C4D1 Predose: number analyzed (Participants) | 1 | 2
  C4D1 Predose | 62.2 (NA) — Standard Deviation was not evaluable as insufficient number of participants. | 364 (77.1)
  C4D1 End of Infusion: number analyzed (Participants) | 1 | 1
  C4D1 End of Infusion | 86.0 (NA) — Standard Deviation was not evaluable as insufficient number of participants. | 595 (NA) — Standard Deviation was not evaluable as insufficient number of participants.

8. Secondary Outcome: Terminal Half-Life (t1/2) of MEDI551
Description: Terminal phase elimination half-life (t1/2) is the time required for half of the drug to be eliminated from the serum.
Time Frame: EOI of Cycle 1 Day 1; Pre-dose and EOI of C1D8, C2D1, C3D1 and C4D1
Population: As-treated Population included all participants who were treated with study drug.
Measure: Mean (Full Range); unit: h
Arm/Group | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg
Number analyzed (Participants) | 5 | 5
h | NA [NA to NA] — t1/2 could not be determined because the participants were not followed for the sufficiently long time. | NA [NA to NA] — t1/2 could not be determined because the participants were not followed for the sufficiently long time.

9. Secondary Outcome: Terminal Half-Life (t1/2) of MEDI0680
Description: Terminal phase elimination half-life (t1/2) is the time required for half of the drug to be eliminated from the serum.
Time Frame: EOI of Cycle 1 Day 2; Pre-dose and EOI of C1D15, C2D1, C3D1 and C4D1
Population: As-treated Population included all participants who were treated with study drug.
Measure: Median (Full Range); unit: h
Arm/Group | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg
Number analyzed (Participants) | 5 | 5
h | NA [NA to NA] — t1/2 could not be determined because the participants were not followed for the sufficiently long time. | NA [NA to NA] — t1/2 could not be determined because the participants were not followed for the sufficiently long time.

10. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) for MEDI-551 and MEDI0680
Description: A participant was considered ADA-positive across the study if they had a positive reading (titer of 50 or higher) at any time point during the study.
Time Frame: 30 min prior to infusion of MEDI-551 on Day 1 of Cycles 1, 2, 6, 9, and 12 and up to 90-days after last dose of study drug (up to approximately 2 years)
Population: As-treated Population included all participants who were treated with study drug.
Measure: Number; unit: Participants
Arm/Group | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg
Number analyzed (Participants) | 5 | 5
Participants | 1 | 0

11. Secondary Outcome: Duration of Complete Response
Description: Duration of Complete Response defined as time from start of first documented Complete Response [CR] to the time of disease progression or death, whichever occurs first. Only participants who have achieved complete response assessed by investigator were evaluated.
Time Frame: From treatment administration to 90-days after last dose of study drug (up to approximately 2 years)
Population: As-treated Population included all participants who were treated with study drug. This parameter was not analyzed as study was discontinued before sufficient data could be collected.
Arm/Group | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Participants With Disease Control
Description: Disease control includes CR (disappearance of all evidence of disease), PR (regression of measurable disease and no new sites), or SD for at least 8 weeks.
Time Frame: From treatment administration to 90-days after last dose of study drug (up to approximately 2 years)
Population: as for outcome 11
Arm/Group | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Duration of Disease Control
Description: Duration of disease control is defined as the time period from the start of disease control event to the event of disease progression.
Time Frame: From treatment administration to 90-days after last dose of study drug (up to approximately 2 years)
Population: as for outcome 11
Arm/Group | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time from the start of study drug administration until the first documentation of disease progression or death due to any cause, whichever occurs first.
Time Frame: From treatment administration to 90-days after last dose of study drug (up to approximately 2 years)
Population: as for outcome 11
Arm/Group | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Overall Survival (OS)
Description: Overall survival defined as the time from the start of study drug administration until death due to any cause.
Time Frame: From treatment administration to 90-days after last dose of study drug (up to approximately 2 years)
Population: as for outcome 11
Arm/Group | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Time to Response (TTR)
Description: Time to response (TTR) defined as the time from the start of study drug administration until the first documentation of disease response. Only participants who have achieved objective response (confirmed CR or confirmed PR) assessed by investigator were evaluated for TTR.
Time Frame: From treatment administration to 90-days after last dose of study drug (up to approximately 2 years)
Population: as for outcome 11
Arm/Group | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From treatment administration to 90 days after last dose of study drug (up to approximately 2 years)
Arm/Group | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 3/5 | 3/5
Serious Adverse Events (participants affected / at risk) | 2/5 | 1/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg (N=5) | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Diffuse large b-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI-551 12 mg/kg and MEDI0680 2.5 mg/kg (N=5) | MEDI-551 12 mg/kg and MEDI0680 10 mg/kg (N=5)
Hypoglobulinaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1)
Chills (General disorders) | 1 (2) | 1 (1)
Fatigue (General disorders) | 2 (3) | 3 (3)
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 2 (5)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (4)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2)
Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (6) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on-going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.